CLINICAL TRIAL: NCT06895148
Title: ADHERE-LPV Advancing Delivery of High-Quality Evidence-Based Respiratory Efforts in Lung-Protective Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ADHERE-LPV
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: This study design allows for comparison of patient outcomes before and after implementation within each hospital while also enabling simultaneous comparisons between hospitals that have and have not yet received the intervention. The cluster randomization approach is necessary, given the order is controlled at the hospital level.
  The intervention will be tested within the MHFV health system which includes a 10-hospital network admitting over 2,500 mechanically ventilated patients annually.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care Ventilator (Active Comparator): Patients in one of the 10 participating hospitals who require mechanical ventilation randomized to the current ventilator order that is used across the health system.
  Interventions: Device: control ventilator
- Experimental Ventilator (Experimental): Patients in one of the 10 participating hospitals who require mechanical ventilation randomized to a new ventilation order
  Interventions: Device: New ventilator

INTERVENTIONS:
Device: New ventilator — The new ventilator order (intervention) was developed using economic behavior theory to decrease the cognitive burden on the ordering provider while enhancing the operability of the order itself. The strategy resulted in a new ventilator order that includes the following changes:
  1. Automatic calculation of the PBW based on the most recent height
  2. If the height is not available, an order to obtain a height will be generated and the choice of tidal volume will be based on cc/kg PBW
  3. Simplify ventilator modes to accurately reflect the standard of care
  4. Reduce duplicative information in the monitoring and comments portion of the order
  5. Cascade ventilator orders based on mode to enhance visualization.
  Arms: Experimental Ventilator
Device: control ventilator — Current ventilator order used by control hospitals
  Arms: Standard of Care Ventilator

SUMMARY:
This study is a cluster randomized trial across 10 hospitals, stratified by hospital size (hospitals with greater than 100 mechanically ventilated patients a year will be classified as large, while those with 100 or fewer will be classified as small). Randomization will occur at the hospital level, ensuring an even distribution of large and small hospitals between study arms. Hospitals assigned to the intervention group will implement an EHR-based strategy designed to enhance adherence to lung-protective ventilation (LPV) for a 9-month intervention period, after which the strategy will be rolled out to all hospitals. The intervention focuses on modifying the ventilator order within the Electronic Health Record (EHR) to encourage default settings aligned with LPV principles. This study design allows for comparison of patient outcomes before and after implementation within each hospital while also enabling simultaneous comparisons between hospitals that have and have not yet received the intervention. The cluster randomization approach is necessary, given the order is controlled at the hospital level.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Requires mechanical ventilation

Exclusion Criteria:

* The patient opted out of research
* The mode ordered does not require a set tidal volume
* Requires ECMO prior to ICU admission
* Data during the use of ECMO
* Hospitalization was for an elective surgery
* The duration of mechanical ventilation was less than 12 hours (these are not the patients that would benefit from LPV)
* Admission code documentation of Do Not Intubate. While rare, in situations where a patient was intubated but whose preferences are contradictory to the current care, mechanical ventilation is managed differently while undergoing goals of care conversations.
* Height was documented as less than 4 feet given the PBW formula was not validated below this height.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1125 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
lung-protective ventilation | 4 hours
  The primary outcome is a binary indicator of lung-protective ventilation (ventilator set at ≤ 8 cc/kg) at the first documented set tidal volume after 4 hours.

SECONDARY OUTCOMES:
Rate (hours) with set tidal volume < 6cc/kg PBW | 72 hours
Rate (hours) exposure to >8 cc/kg PBW | 72 hours
Rate (hours) exposure to >10 cc/kg PBW | 72 hours
Time to adhere to ≤ 8 cc/kg per day: Of all patients set to >8 cc/kg per day, how long did it take for the patient to receive ≤ 8 cc/kg per day? | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States